CLINICAL TRIAL: NCT03268850
Title: Living Donor Lost Wages Trial
Brief Title: Living Kidney Donor Lost Wages Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, James Rodrigue, Primary Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2017P000213
Record Dates: First submitted 2017-08-22; First posted 2017-08-31 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Kidney Diseases
Keywords: LDKT; Live donor transplantation; Kidney transplantation
MeSH Terms: conditions — Kidney Diseases | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Candidates will be randomized 1:1 to the LW-A or LW-B arm, with stratification for race. The investigators will prepare the randomization schedule using permuted blocks of randomly varying size to limit predictability and imbalances in arm assignment throughout the study. KT candidates will be informed of group assignment immediately after consenting to the study.
Who Masked: Care Provider, Investigator
Masking Description: Allocation will be concealed from the study investigators; however, research assistants conducting the assessments will not be blinded since the assessment protocol differs based on group assignment. Study participants will know which arm they are in, but not the reimbursement amount of the other arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LW-A (Experimental): The Lost Wages A (LW-A) arm will be composed of kidney transplant patients meeting the inclusion criteria. This arm allows for possible wage reimbursement of living donor lost wages up to a certain amount. This will also include standard of care.
  Interventions: Other: Standard of Care; Behavioral: Wage Reimbursement A
- LW-B (Experimental): The Lost Wages B (LW-B) arm will be composed of kidney transplant patients meeting the inclusion criteria. This arm allows for possible wage reimbursement of living donor lost wages up to a different amount. This will also include standard of care.
  Interventions: Other: Standard of Care; Behavioral: Wage Reimbursement B

INTERVENTIONS:
Other: Standard of Care — All patients participating in the study will continue to receive usual care. Kidney transplant (KT) candidates are advised that live donor kidney transplantation (LDKT) is their best treatment option and are encouraged to initiate living donor (LD) discussions with family members and friends.
Behavioral: Wage Reimbursement A — Enrolled KT candidates will be informed that, in addition to the National Living Donor Assistance Center (NLDAC) program, their LD may be eligible to receive reimbursement for wages lost during the donation recovery period - up to a certain amount, based on randomization. They will be given information describing the LW program, eligibility criteria, and application process to share with potential LDs. At the time of study enrollment, KT candidates will consent to the LD nurse coordinator informing all of their potential LDs about the study and the potential for reimbursement of LD lost wages.
  Reimbursement will occur for those LDs who file an application, provide the required documentation, and meet eligibility criteria.
  Arms: LW-A
Behavioral: Wage Reimbursement B — Enrolled KT candidates will be informed that, in addition to the National Living Donor Assistance Center (NLDAC) program, their LD may be eligible to receive reimbursement for wages lost during the donation recovery period - up to a certain amount (different from LW-A), based on randomization. They will be given information describing the LW program, eligibility criteria, and application process to share with potential LDs. At the time of study enrollment, KT candidates will consent to the LD nurse coordinator informing all of their potential LDs about the study and the potential for reimbursement of LD lost wages.
  Reimbursement will occur for those LDs who file an application, provide the required documentation, and meet eligibility criteria.
  Arms: LW-B

SUMMARY:
This study aims to evaluate the effectiveness of offering reimbursement for living donor lost wages on the rate of live donor kidney transplantation.

DETAILED DESCRIPTION:
Live donor kidney transplantation (LDKT) accelerates the path to transplantation and yields superior outcomes compared to dialysis and deceased donor kidney transplantation (KT). However, the annual number of LDKTs has declined over the last decade, particularly among minority and low-income patients. The investigators hypothesize, and have preliminary data to support, that the financial impact on living donors (LDs) is a major contributor to the LDKT decline and for persistent racial disparities in LDKT rates. Many LDs have substantial non-reimbursed direct and indirect costs, most notably the loss of income or wages following surgery. In this study, the investigators will: (1) evaluate the effectiveness of offering reimbursement for LD lost wages on the LDKT rate; (2) examine whether offering reimbursement for LD lost wages reduces known racial disparities in LDKT; and (3) determine whether study outcomes differ significantly by maximum reimbursement amount for LD lost wages.

ELIGIBILITY:
Inclusion Criteria:

* For KT patients:
* Chronic Kidney Disease (CKD) stage 4/5
* Approved for kidney transplant (KT) listing or active on KT waiting list
* For patients listed at multiple centers: primary listing at Beth Israel Deaconess Medical Center (BIDMC)
* For LDs:
* Their KT candidate is enrolled in the trial

Exclusion Criteria:

* For KT patients:
* KT candidate has a potential LD approved, with surgery scheduled
* Listed for multi-organ transplantation
* Temporarily unavailable (TU) status on KT waiting list
* Current enrollment in another study to increase LDKT likelihood
* For LDs:
* Not residing in the US

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of wage reimbursement on LDKT rate | 1 year
  LDKT rate in KT candidates compared to historical matched control group
Effect of wage reimbursement on racial disparities in LDKT | 1 year
  LDKT rate among minorities
Difference between reimbursement arms | 1 year
  LDKT rate in KT candidates in LW-A arm as compared to LDKT rate in KT candidates in LW-B arm

CONTACTS AND LOCATIONS:
Locations (1):
- BIDMC Transplant Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No